CLINICAL TRIAL: NCT03948932
Title: Cervical "Resistance" Measurements - a Novel Method for Evaluation of Cervical "Ripeness" Prior to Labor Induction
Brief Title: Cervix Uteri "Resistance" Measurements
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, ROY LAUTERBACH MD, Principal Investigator, Rambam Health Care Campus
Other Study IDs: 0246-16-RMB
Record Dates: First submitted 2019-05-08; First posted 2019-05-14 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Induction of Labor Affected Fetus / Newborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Transvaginal sonography — Measurement of cervical length via transvaginal sonography prior to labor induction.
Device: Pressure watch — Measurement of inflation pressure in a cervical ripening balloon is PSI units.

SUMMARY:
Pregnant women at term, after 37 weeks' gestation will undergo cervical ripening for labor induction via cervical ripening balloon. Transvaginal sonography will be performed before balloon insertion. During balloon insertion and after uterine balloon inflation a pressure watch will be attached to the balloon and inflation pressures of the vaginal balloon will be measured and documented.

DETAILED DESCRIPTION:
The investigators routinely use the Cook balloon catheter 13 for mechanical induction of labor 10-11 - this is a medical grade, double balloon catheter, comprised of a slender, flexible tube open at one end and closed at the opposite end; an inflatable distal balloon fixed to the tube at its closed end and designed to be inflated in the uterus; an inflatable proximal balloon located slightly below the uterine balloon (labeled as the cervical balloon).

The catheter will be inserted according to the manufacturer's instructions with the patient in a lithotomy position under visualization of the cervix. When both balloons are inserted, the uterine balloon will be inflated through valve V1; using 40 ml of sterile saline solution. With a slight downward pull on the catheter, the cervical balloon will be located inside the cervix. In order to measure the cervical resistance, the investigators will connect a sensitive, passive pressure gauge to the cervical inflated balloon with the use of a by a bi-directional valve. At this point the investigators will gradually inflate the cervical balloon via valve V2 with 80 ml of sterile saline solution. The cervical resistance will be measured and documented every 10 ml. Finally, the uterine balloon will be further inflated with additional saline to a volume of 40 ml. (as per our standard mechanical induction protocol). The investigators believe that this system provides an objective and quantifiable evaluation of the pressure exerted on the cervical balloon as it is gradually inflated. As the cervical stiffness ("resistance") increases the pressure within the cervical balloon will be higher with a given volume of fluid within it. Therefore, the investigators define cervical resistance as the pressure vs. volume curve within the cervical balloon.

A group of 100 patients, (50 multiparas & 50 nulliparas) with an obstetrical or medical indication for induction of labor will be recruited and consented for participation in this study. A transvaginal ultrasound will be performed prior to the initiation of the procedure to exclude placenta previa and to confirm a vertex presentation. Cervical length and angle will be recorded. All women will undergo a pelvic examination in order to obtain an initial Bishop Score.

ELIGIBILITY:
Inclusion Criteria:

* Obstetrical or medical indication for induction of labor
* Unfavorable cervix
* Gestational age between 24 - 42 weeks
* Singleton pregnancy

Exclusion Criteria:

* Any contraindication for vaginal delivery
* Rupture of membranes
* Fetal malformations incompatible with life
* Amnionitis
* Genital viral infection (HIV, HCV, HBV)

Ages: 18 Years to 44 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: Pregnant women between 24-42 weeks gestation that are candidates for labor induction with a cervical ripening balloon.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Volume versus pressure | From patient admission up to 24 hours postpartum.
  To define pressure versus volume characteristics of the expanding uterine cervical balloon.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Lauterbach, MD, Principal Investigator — Rambam healthcare campus
Locations (1):
- Rambam health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No